CLINICAL TRIAL: NCT00099554
Title: A Phase 4, Open-Label, Single Arm, Observational Study Evaluating the Effectiveness and Safety of Enbrel® (Etanercept) 50 mg Once Weekly in Rheumatoid Arthritis Subjects Who Have Failed Remicade® (Infliximab)
Brief Title: Effectiveness and Safety of Enbrel® (Etanercept) in Rheumatoid Arthritis Subjects Who Have Failed Remicade® (Infliximab)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20030236
Record Dates: First submitted 2004-12-16; First posted 2004-12-17 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

INTERVENTIONS:
Drug: Etanercept

SUMMARY:
The purpose of this study is to evaluate the proportion of Rheumatoid Arthritis (RA) subjects achieving a "good" or "moderate" DAS28 response (EULAR28 criteria) at Week 16 with etanercept 50 mg subcutaneously (SC) once weekly in patients who have failed infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Adults with RA (ACR criteria) for greater than or equal to 6 months
* Infliximab treatment for at least 18 weeks
* Infliximab infusion prior to screening at an increased dosing regimen: 5 mg/kg every 4-8 weeks (dose), OR, 3 mg/kg every 4-6 weeks (frequency)
* Failing infliximab defined by ALL of the following at screening and baseline visit: Disease Activity Score (DAS 28) greater than or equal to 4.5, greater than or equal to 5 swollen joints, greater than or equal to 5 tender joints
* Subjects must be receiving stable methotrexate (MTX), at a dose of greater than or equal to 10 mg/week at least 10 weeks prior to screening
* Stable disease modifying anti-rheumatic drugs (DMARD) therapy (including sulfasalazine, hydroxychloroquine), greater than or equal to 8 weeks prior to screening
* Stable dose corticosteroids, less than 10 mg/day at greater than or equal to 4 weeks prior to screening
* Stable dose of non-steroidal anti-inflammatory drugs (NSAIDs) greater than or equal to 1 week prior to screening

Exclusion Criteria:

* ACR functional class IV - Prior treatment with etanercept
* Receipt of any investigational drug/biologic within 28 days of study drug initiation
* Active infection or predisposition to infection
* Elective surgery planned during study period
* Intra-articular, soft tissue, or intramuscular corticosteroid injections during 4 weeks prior to screening
* Contraindications to etanercept as defined in the package insert
* Severe co-morbidities: History of cancer within 5 years; Diagnosis of class III or IV congestive heart failure (CHF); Uncontrolled hypertension (HTN); CNS-demyelinating events suggestive of multiple sclerosis (MS); Known HIV-positive status; Oxygen-dependent pulmonary status; Chronic hepatitis B or C; Systemic Lupus Erythematosus (SLE); Active or prior history of tuberculosis (TB) (or known exposure) or positive PPD without adequate TB prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-05

PRIMARY OUTCOMES:
Proportion of subjects achieving a "good" or "moderate" DAS28 response (as defined by EULAR28 criteria) at Week 16.

SECONDARY OUTCOMES:
Proportion of subjects who achieve ACR 20, 50, and 70 responses at Weeks 8 and 16.
Proportion of subjects who achieve good or moderate DAS28 response at Week 8 and the proportion who achieve remission (DAS28 less than 2.6) at Weeks 8 and 16
Absolute and percent changes from baseline in components of the ACR and DAS28 criteria (including HAQ) at Weeks 8 and 16.
Absolute changes from baseline in SF-36 and Valued Life Activities at Weeks 8 and 16
Subject incidence rate of SAEs over 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Bingham CO 3rd, Ince A, Haraoui B, Keystone EC, Chon Y, Baumgartner S. Effectiveness and safety of etanercept in subjects with RA who have failed infliximab therapy: 16-week, open-label, observational study. Curr Med Res Opin. 2009 May;25(5):1131-42. doi: 10.1185/03007990902841010. PMID 19317607
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20030236.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/